CLINICAL TRIAL: NCT01021293
Title: Immunogenicity and Safety of GSK Biologicals' IPV (Poliorix™) in Infants
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline Biologicals' Poliorix™ Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112679; 2011-003167-30 (EudraCT Number)
Record Dates: First submitted 2009-11-25; First posted 2009-11-26 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Poliomyelitis; Poliomyelitis Vaccines
Keywords: Poliorix; IPV
MeSH Terms: conditions — Poliomyelitis | interventions — Poliovirus Vaccine, Oral

ARMS (2):
- Poliorix Group (Experimental): Healthy male and female Chinese infants between, and including 60 and 90 days of age, who received 3 doses of Poliorix™ (IPV) vaccine at 2, 3 and 4 months of age, administered intramuscularly into the anterolateral side of the right thigh.
  Interventions: Biological: Poliorix™
- Control Group (Active Comparator): Healthy male and female Chinese infants between, and including 60 and 90 days of age, who received 3 doses of Oral Poliomyelitis Vaccine (OPV) at 2, 3 and 4 months of age, according to the vaccination policy recommended in China.
  Interventions: Biological: Oral Poliovirus vaccine

INTERVENTIONS:
Biological: Poliorix™ — 3 doses, intramuscular administration
  Arms: Poliorix Group
Biological: Oral Poliovirus vaccine — 3 doses, oral administration
  Arms: Control Group

SUMMARY:
The purpose of the study is to evaluate the immunogenicity and safety of Poliorix™ when administered to healthy Chinese infants at 2, 3 and 4 months of age.

ELIGIBILITY:
Inclusion Criteria:

* A male or female infant between, and including, 60 and 90 days of age at the time of the first vaccination.
* Born after a gestation period of 36 to 42 weeks inclusive.
* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative (LAR) (s) can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to vaccination, or planned administration during the study period, with exception of DTP, Hib and/or hepatitis B vaccine(s).
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Evidence of previous or intercurrent poliomyelitis disease or vaccination.
* History of seizures or progressive neurological disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness.
* Child in care.

The following condition is temporary or self-limiting, and a subject may be vaccinated once the condition has resolved and if no other exclusion criteria are met:

• Current febrile illness or axillary temperature > 37.0 ºC or other moderate to severe illness within 24 hours of study vaccine administration.

Ages: 60 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1101 (Actual)
Dates: Start 2009-11-28 (Actual); Primary Completion 2010-07-05 (Actual); Study Completion 2010-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wuzhou, Guangxi, China

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=268

REFERENCES:
- [Background] Li R et al. Immunogenicity and safety of an inactivated poliovirus vaccine in Chinese infants. Abstract presented at the 7th World Congress for World Society for Pediatric Infectious Diseases (WSPID). The Melbourne, The Australia, 16-19 November 2011.
- [Background] Li R, Li CG, Li Y, Liu Y, Zhao H, Chen X, Kuriyakose S, Van Der Meeren O, Hardt K, Hezareh M, Roy-Ghanta S. Primary and booster vaccination with an inactivated poliovirus vaccine (IPV) is immunogenic and well-tolerated in infants and toddlers in China. Vaccine. 2016 Mar 14;34(12):1436-43. doi: 10.1016/j.vaccine.2016.02.010. Epub 2016 Feb 9. PMID 26873055
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 112679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 1101 enrolled subjects, one subject was not randomised and administered any vaccine as the parents of the subject refused to vaccinate their child after blood collection at Visit 1 and withdrew their consent.
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Poliorix Group: Healthy male and female Chinese infants between, and including 60 and 90 days of age, who received 3 doses of Poliorix (IPV) vaccine at 2, 3 and 4 months of age, administered intramuscularly into the anterolateral side of the right thigh.
Period: Overall Study
Arm/Group | Poliorix Group | Control Group
Started | 550 | 550
Completed | 538 | 526
Not Completed | 12 | 24
Not completed — Serious Adverse Event | 2 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Migrated/moved from study area | 6 | 18
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Poliorix Group | Control Group | Total
Number analyzed (Participants) | 550 | 550 | 1100
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 10 (1.16) | 10.1 (1.18) | 10.05 (1.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 268 | 259 | 527
  Male | 282 | 291 | 573
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-Chinese heritage | 550 | 550 | 1100

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects Against Poliovirus Types 1, 2 and 3
Description: A seroprotected subject was defined as a vaccinated subject with anti-polio types 1, 2 and 3 titers greater than or equal to (≥) 8 effective dose 50 (ED50).
Time Frame: At Month 3, one month after the third vaccine dose
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome variables and assay results for antibodies against at least one study vaccine antigen component after vaccination were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Poliorix Group | Control Group
Number analyzed (Participants) | 306 | 296
Participants
  Anti-poliovirus 1 | 306 | 296
  Anti-poliovirus 2 | 306 | 296
  Anti-poliovirus 3 | 306 | 291
Statistical Analysis 1: Comparison: Poliorix Group vs Control Group; Non-inferiority of Poliorix™ as compared to OPV; Test type: Non-Inferiority — Non-inferiority of Poliorix™ vaccine as compared to OPV vaccine in terms of the immune response to poliovirus type 1 one month after the third vaccine dose. Non-inferiority in terms of immunogenicity to poliovirus antigens was demonstrated if the upper limit of the 95% confidence interval (CI) on the group difference [Control Group minus Poliorix Group] in the percentage of seroprotected subjects; Difference in seroprotection rate = 0, 95% CI 2-sided [-1.28 to 1.24]
Statistical Analysis 2: Comparison: Poliorix Group vs Control Group; Non-inferiority of Poliorix™ as compared to OPV; Test type: Non-Inferiority — Non-inferiority of Poliorix™ vaccine as compared to OPV vaccine in terms of the immune response to poliovirus type 2 one month after the third vaccine dose. Non-inferiority in terms of immunogenicity to poliovirus antigens was demonstrated if the upper limit of the 95% confidence interval (CI) on the group difference [Control Group minus Poliorix Group] in the percentage of seroprotected subjects; Difference in seroprotection rate = 0, 95% CI 2-sided [-1.28 to 1.24]
Statistical Analysis 3: Comparison: Poliorix Group vs Control Group; Non-inferiority of Poliorix™ as compared to OPV; Test type: Non-Inferiority — Non-inferiority of Poliorix™ vaccine as compared to OPV vaccine in terms of the immune response to poliovirus type 3 one month after the third vaccine dose. Non-inferiority in terms of immunogenicity to poliovirus antigens was demonstrated if the upper limit of the 95% confidence interval (CI) on the group difference [Control Group minus Poliorix Group] in the percentage of seroprotected subjects; Difference in seroprotection rate = -1.69, 95% CI 2-sided [-3.9 to -0.44]

2. Secondary Outcome: Number of Seroprotected Subjects Against Poliovirus Types 1, 2 and 3
Description: A seroprotected subject was defined as a vaccinated subject with anti-poliovirus types 1, 2 and 3 titers ≥ 8 ED50.
Time Frame: At Day 0, prior to the first vaccine dose
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome variables and assay results for antibodies against at least one study vaccine antigen component after vaccination were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Poliorix Group | Control Group
Number analyzed (Participants) | 306 | 296
Participants
  Anti-poliovirus 1 | 131 | 113
  Anti-poliovirus 2 | 93 | 99
  Anti-poliovirus 3 | 48 | 52

3. Secondary Outcome: Anti-poliovirus Types 1, 2 and 3 Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: Prior to the first vaccine dose (Day 0) and one month after the third vaccine dose (Month 3)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Poliorix Group | Control Group
Number analyzed (Participants) | 306 | 296
Titers
  Anti-poliovirus 1, D0 | 8.7 [7.6 to 9.8] | 7.8 [6.9 to 8.9]
  Anti-poliovirus 1, M3 | 485.1 [436.7 to 538.9] | 2817 [2479.5 to 3200.4]
  Anti-poliovirus 2, D0 | 6.5 [5.9 to 7.1] | 7.2 [6.5 to 8.1]
  Anti-poliovirus 2, M3 | 234.3 [209 to 262.6] | 468.5 [416.6 to 526.9]
  Anti-poliovirus 3, D0 | 5.2 [4.8 to 5.7] | 5.2 [4.8 to 5.7]
  Anti-poliovirus 3, M3 | 824.3 [725.3 to 936.9] | 423.4 [363.3 to 493.3]

4. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of any local symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimeters (mm) of injection site. This outcome measure concerns subjects from the Poliorix Group only.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following each vaccine dose and across doses
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented, who had filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | Poliorix Group
Number analyzed (Participants) | 550
Participants
  Any Pain, Dose 1 | 80
  Grade 3 Pain, Dose 1 | 1
  Any Redness, Dose 1 | 20
  Grade 3 Redness, Dose 1 | 0
  Any Swelling, Dose 1 | 9
  Grade 3 Swelling, Dose 1 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 543
  Any Pain, Dose 2 | 58
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 543
  Grade 3 Pain, Dose 2 | 2
  Any Redness, Dose 2: number analyzed (Participants) | 543
  Any Redness, Dose 2 | 23
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 543
  Grade 3 Redness, Dose 2 | 1
  Any Swelling, Dose 2: number analyzed (Participants) | 543
  Any Swelling, Dose 2 | 8
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 543
  Grade 3 Swelling, Dose 2 | 1
  Any Pain, Dose 3: number analyzed (Participants) | 540
  Any Pain, Dose 3 | 41
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 540
  Grade 3 Pain, Dose 3 | 0
  Any Redness, Dose 3: number analyzed (Participants) | 540
  Any Redness, Dose 3 | 15
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 540
  Grade 3 Redness, Dose 3 | 0
  Any Swelling, Dose 3: number analyzed (Participants) | 540
  Any Swelling, Dose 3 | 6
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 540
  Grade 3 Swelling, Dose 3 | 0
  Any Pain, Across doses | 113
  Grade 3 Pain, Across doses | 3
  Any Redness, Across doses | 46
  Grade 3 Redness, Across doses | 1
  Any Swelling, Across doses | 18
  Grade 3 Swelling, Across doses | 1

5. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, gastrointestinal symptoms, irritability/fussiness, loss of appetite and fever [defined as axillary temperature higher than (>) 37.0°C degrees Celsius]. Gastrointestinal symptoms included nausea, vomiting, diarrhoea and/or abdominal pain. Any = occurrence of any general symptom regardless of intensity grade or relationship to vaccination. Grade 3 drowsiness = drowsiness that prevented normal activity. Grade 3 irritability = crying that could not be comforted/ prevented normal activity. Grade 3 loss of appetite = subject did not eat at all. Grade 3 gastrointestinal symptoms = gastrointestinal symptoms that prevented normal activity. Grade 3 fever= temperature > 39°C. Related = symptom assessed by the investigator as causally related to the vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following each vaccine dose and across doses
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Poliorix Group | Control Group
Number analyzed (Participants) | 550 | 550
Participants
  Any Drowsiness, Dose 1 | 99 | 75
  Grade 3 Drowsiness, Dose 1 | 0 | 1
  Related Drowsiness, Dose 1 | 71 | 51
  Any Gastrointestinal Symptoms, Dose 1 | 102 | 89
  Grade 3 Gastrointestinal, Dose 1 | 0 | 2
  Related Gastrointestinal, Dose 1 | 44 | 43
  Any Irritability/Fussiness, Dose 1 | 160 | 151
  Grade 3 Irritability/Fussiness, Dose 1 | 1 | 5
  Related Irritability/Fussiness, Dose 1 | 130 | 105
  Any Loss of appetite, Dose 1 | 82 | 83
  Grade 3 Loss of appetite, Dose 1 | 0 | 1
  Related Loss of appetite, Dose 1 | 54 | 47
  Any temperature, Dose 1 | 39 | 20
  Grade 3 temperature, Dose 1 | 0 | 0
  Related temperature, Dose 1 | 28 | 10
  Any Drowsiness, Dose 2: number analyzed (Participants) | 543 | 544
  Any Drowsiness, Dose 2 | 68 | 50
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 543 | 544
  Grade 3 Drowsiness, Dose 2 | 2 | 0
  Related Drowsiness, Dose 2: number analyzed (Participants) | 543 | 544
  Related Drowsiness, Dose 2 | 51 | 25
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 543 | 544
  Any Gastrointestinal, Dose 2 | 66 | 67
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 543 | 544
  Grade 3 Gastrointestinal, Dose 2 | 2 | 1
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 543 | 544
  Related Gastrointestinal, Dose 2 | 32 | 35
  Any Irritability/Fussiness, Dose 2: number analyzed (Participants) | 543 | 544
  Any Irritability/Fussiness, Dose 2 | 121 | 86
  Grade 3 Irritability/Fussiness, Dose 2: number analyzed (Participants) | 543 | 544
  Grade 3 Irritability/Fussiness, Dose 2 | 7 | 2
  Related Irritability/Fussiness, Dose 2: number analyzed (Participants) | 543 | 544
  Related Irritability/Fussiness, Dose 2 | 105 | 50
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 543 | 544
  Any Loss of appetite, Dose 2 | 70 | 78
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 543 | 544
  Grade 3 Loss of appetite, Dose 2 | 3 | 0
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 543 | 544
  Related Loss of appetite, Dose 2 | 48 | 47
  Any temperature, Dose 2: number analyzed (Participants) | 543 | 544
  Any temperature, Dose 2 | 39 | 26
  Grade 3 temperature, Dose 2: number analyzed (Participants) | 543 | 544
  Grade 3 temperature, Dose 2 | 2 | 1
  Related temperature, Dose 2: number analyzed (Participants) | 543 | 544
  Related temperature, Dose 2 | 29 | 11
  Any Drowsiness, Dose 3: number analyzed (Participants) | 540 | 534
  Any Drowsiness, Dose 3 | 47 | 45
  Grade 3 Drowsiness, Dose 3: number analyzed (Participants) | 540 | 534
  Grade 3 Drowsiness, Dose 3 | 2 | 1
  Related Drowsiness, Dose 3: number analyzed (Participants) | 540 | 534
  Related Drowsiness, Dose 3 | 36 | 25
  Any Gastrointestinal, Dose 3: number analyzed (Participants) | 540 | 534
  Any Gastrointestinal, Dose 3 | 46 | 67
  Grade 3 Gastrointestinal, Dose 3: number analyzed (Participants) | 540 | 534
  Grade 3 Gastrointestinal, Dose 3 | 3 | 0
  Related Gastrointestinal, Dose 3: number analyzed (Participants) | 540 | 534
  Related Gastrointestinal, Dose 3 | 16 | 25
  Any Irritability/Fussiness, Dose 3: number analyzed (Participants) | 540 | 534
  Any Irritability/Fussiness, Dose 3 | 87 | 72
  Grade 3 Irritability/Fussiness, Dose 3: number analyzed (Participants) | 540 | 534
  Grade 3 Irritability/Fussiness, Dose 3 | 2 | 2
  Related Irritability/Fussiness, Dose 3: number analyzed (Participants) | 540 | 534
  Related Irritability/Fussiness, Dose 3 | 77 | 44
  Any Loss of appetite, Dose 3: number analyzed (Participants) | 540 | 534
  Any Loss of appetite, Dose 3 | 52 | 64
  Grade 3 Loss of appetite, Dose 3: number analyzed (Participants) | 540 | 534
  Grade 3 Loss of appetite, Dose 3 | 0 | 0
  Related Loss of appetite, Dose 3: number analyzed (Participants) | 540 | 534
  Related Loss of appetite, Dose 3 | 34 | 36
  Any temperature, Dose 3: number analyzed (Participants) | 540 | 534
  Any temperature, Dose 3 | 33 | 32
  Grade 3 temperature, Dose 3: number analyzed (Participants) | 540 | 534
  Grade 3 temperature, Dose 3 | 0 | 2
  Related temperature, Dose 3: number analyzed (Participants) | 540 | 534
  Related temperature, Dose 3 | 18 | 17
  Any Drowsiness, Across doses | 140 | 125
  Grade 3 Drowsiness, Across doses | 4 | 2
  Related Drowsiness, Across doses | 115 | 80
  Any Gastrointestinal, Across doses | 154 | 156
  Grade 3 Gastrointestinal, Across doses | 5 | 3
  Related Gastrointestinal, Across doses | 76 | 87
  Any Irritability, Across doses | 244 | 216
  Grade 3 Irritability, Across doses | 10 | 9
  Related Irritability, Across doses | 214 | 159
  Any Loss of appetite, Across doses | 147 | 168
  Grade 3 Loss of appetite, Across doses | 3 | 1
  Related Loss of appetite, Across doses | 109 | 109
  Any Fever, Across doses | 99 | 71
  Grade 3 Fever, Across doses | 2 | 3
  Related Fever, Across doses | 68 | 36

6. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within the 31-day (Days 0-30) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Poliorix Group | Control Group
Number analyzed (Participants) | 550 | 550
Participants | 155 | 162

7. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity.
Time Frame: During the entire study period (from Day 0 to Month 3)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Groups:
- Control Group: Healthy male and female Chinese infants between, and including 60 and 90 days of age, who received 3 doses of Oral Poliomyelitis Vaccine (OPV) vaccine at 2, 3 and 4 months of age, according to the vaccination policy recommended in China.
Arm/Group | Poliorix Group | Control Group
Number analyzed (Participants) | 550 | 550
Participants | 3 | 6

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Days 0-3) post-vaccination period. Unsolicited AEs: within the 31-day (Days 0-30) post-vaccination period. SAEs: during the entire study period (from Day 0 up to Month 3).
Arm/Group | Poliorix Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/550 | 0/550
Serious Adverse Events (participants affected / at risk) | 3/550 | 6/550
Other Adverse Events (participants affected / at risk) | 391/550 | 366/550
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Poliorix Group (N=550) | Control Group (N=550)
Cardiac failure (Cardiac disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Poliorix Group (N=550) | Control Group (N=550)
Upper respiratory tract infection (Infections and infestations) | 99 | 97
Nasopharyngitis (Infections and infestations) | 32 | 38
Pain (General disorders) | 113 | 0
Redness (General disorders) | 46 | 0
Drowsiness (General disorders) | 140 | 125
Gastrointestinal symptoms (General disorders) | 154 | 156
Irritability/Fussiness (General disorders) | 244 | 216
Loss of appetite (General disorders) | 147 | 168
Fever (Axillary) (General disorders) | 99 | 71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.